CLINICAL TRIAL: NCT07160296
Title: Supporting Treatment Resilience With Optimized Nutrition and Guided Exercise in Head and Neck Cancer Patients Undergoing Chemoradiation
Acronym: STRONGER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Renown Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1002504325
Record Dates: First submitted 2025-08-14; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Cancer
Keywords: ChemoRT; HNC; Wellness
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open Label Arm (Experimental): Participate in a 20-week lifestyle program that includes:
  * Nutrition counseling: Weekly group sessions with an oncology dietitian, including individualized calorie and protein goals.
  * Exercise: Home-based resistance and mobility exercises twice per week using online videos, and daily walking with self-tracking.
  * Wellness education: Weekly group sessions focused on stress management, sleep, fatigue, and mindset, facilitated by a health and wellness coach. Five of the 20 sessions will include a Speech, Voice, Swallowing, and Airway Care in Head & Neck Cancer training series led by a speech pathologist.
  Interventions: Behavioral: 20-Week Lifestyle Program

INTERVENTIONS:
Behavioral: 20-Week Lifestyle Program — Nutrition counseling: Weekly group sessions with an oncology dietitian, including individualized calorie and protein goals.
  Exercise: Home-based resistance and mobility exercises twice per week using online videos, and daily walking with self-tracking.
  Wellness education: Weekly group sessions focused on stress management, sleep, fatigue, and mindset, facilitated by a health and wellness coach. Five of the 20 sessions will include a Speech, Voice, Swallowing, and Airway Care in Head & Neck Cancer training series led by a speech pathologist.

SUMMARY:
The purpose of this study to find out whether a structured lifestyle intervention-combining nutrition counseling, guided exercise, and wellness education-can help reduce treatment-related side effects and improve physical function, resilience, and quality of life in patients with head and neck cancer undergoing chemoradiation therapy (chemoRT).

Benefits of research cannot be guaranteed but we hope to learn whether this intervention is feasible and acceptable during active cancer treatment, and whether it can help preserve lean body mass, improve strength and endurance, and support emotional well-being. The findings will inform the design of a future larger clinical trial.

DETAILED DESCRIPTION:
This pilot study aims to assess the feasibility and preliminary effects of a multimodal lifestyle intervention-integrating nutrition optimization, guided exercise, and wellness education-on sarcopenia and resilience during treatment for HNC. The scope of these assessments are not experimental in nature, but will be applied in combination for this patient population as supplemental care. While the interventions are not uncommon for cancer patients, particularly as cancer patients may seek these care options independently during treatment, the participants will not be billed for these services as they are experimental in that they are not in standard treatment guidelines.

This pilot study will inform the refinement of the STRONGER intervention for future use in a larger randomized controlled trial. It will test implementation logistics and provide preliminary data on intervention benefits for patients undergoing intensive cancer therapy, such as chemoRT.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years old with biopsy-confirmed squamous cell carcinoma of the head and neck
* Planned for definitive or adjuvant chemoRT
* ECOG performance status 0-2
* Ability to participate in light-to-moderate physical activity
* Able to provide informed consent

Exclusion Criteria:

* Severe malnutrition requiring exclusive enteral feeding at baseline
* Comorbidities that preclude safe participation in exercise
* Cognitive or psychiatric conditions that impair study engagement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Program: Recruitment Rate | From enrollment to the end of the intervention at 20 weeks
  Percentage of eligible patients who enroll in the study. Unit of Measure: Percentage (%) enrolled compared to not enrolled of eligible participants approached.
Program Acceptability | From enrollment to the end of the intervention at 20 weeks
  A five-point Likert Scale and open-ended prompts will be used to assess acceptability (see appendix) upon completion of the 20-week intervention
Feasibility of Program: Retention Rate | From enrollment to 20 weeks
  Percentage of enrolled participants who complete the 20-week intervention. Unit of Measure: Percentage (%) of participants who complete the program
Feasibility of Program: Session Attendance | Over the 20-week intervention period
  Number of nutrition and wellness group sessions attended per participant. Unit of Measure: Count (number of sessions attended)
Feasibility of Program: Adherence to Exercise Plan - Resistance Training | Over the 20-week intervention period
  Percentage of prescribed resistance training sessions (2x/week) completed by each participant.
  Unit of Measure: Percentage (%) completion rate
Feasibility of Program: Adherence to Exercise Plan - Walking Goals | Over the 20-week intervention period
  Percentage of weekly walking goals met by each participant. Unit of Measure: Percentage (%) completed goals
Feasibility of Program: Data Completeness | From baseline to 20-week follow-up
  Percentage of participants with complete data at baseline, end of treatment, and 20-week follow-up.
  Unit of Measure: Percentage (%) complete data
Feasibility of Program: Protocol Fidelity | Over the 20-week intervention period
  Percentage of intervention components delivered as intended, per protocol. Unit of Measure: Percentage (%) delivered
Feasibility of Program: Adverse Events | Over the 20-week intervention period
  Number of safety issues reported by staff or participants during the intervention.
  Unit of Measure: Count (number of adverse events)

SECONDARY OUTCOMES:
Clinical Outcomes of Interest: Quality of Life | From enrollment to the end of the intervention at 20 weeks
  Assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) at baseline and week 20.
  Unit of Measure: Units on a scale (0-100) Interpretation: Higher scores indicate better functioning or quality of life for functional scales; higher scores indicate worse symptoms for symptom scales.
Clinical Outcomes of Interest: Change in Sarcopenia Risk | From baseline to week 20
  Assessed using the SARC-F Questionnaire at baseline and week 20. Unit of Measure: Units on a scale (0-10) Interpretation: Higher scores indicate greater risk of sarcopenia.
Clinical Outcomes of Interest: Change in Depression Symptoms | From baseline to week 20
  Assessed using the Patient Health Questionnaire-9 (PHQ-9) at baseline and week 20.
  Unit of Measure: Units on a scale (0-27) Interpretation: Higher scores indicate more severe depressive symptoms.
Clinical Outcomes of Interest: Change in Anxiety Symptoms | From baseline to week 20
  Assessed using the Generalized Anxiety Disorder 7-item scale (GAD-7) at baseline and week 20.
  Unit of Measure: Units on a scale (0-21) Interpretation: Higher scores indicate more severe anxiety symptoms.
Clinical Outcomes of Interest: Change in Lean Body Mass | From baseline to week 20
  Measured via bioimpedance scale at baseline, week 7, and week 20. Unit of Measure: Kilograms (kg)
Clinical Outcomes of Interest: Change in Body Weight | From baseline to week 20
  Measured at baseline, bi-weekly, and week 20. Unit of Measure: Kilograms (kg)
Clinical Outcomes of Interest: Change in Grip Strength | From baseline to week 20
  Measured using a hand dynamometer at baseline, week 7, and week 20. Unit of Measure: Kilograms (kg)
Clinical Outcomes of Interest: Change in Functional Capacity (6MWT) | From baseline to week 20
  Measured using the 6-minute walk test at baseline, week 7, and week 20. Unit of Measure: Meters walked

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Renown Regional Medical Center, Reno, Nevada
  - Conrad Breast Center at South Meadows, Reno, Nevada

IPD SHARING:
Plan to Share IPD: Undecided